CLINICAL TRIAL: NCT02581072
Title: A Double-blind, Double-dummy, Randomized, 4-period Crossover Study to Define the ECG Effects of SB204 Using a Clinical and Supratherapeutic Dose Compared With Placebo and Moxifloxacin in Subjects With Acne Vulgaris: A Thorough ECG STudy
Brief Title: A Thorough ECG Study in Subjects With Acne Vulgaris Treated With SB204
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC104
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SB204 4% (Experimental): SB204 4% once
  Interventions: Drug: SB204 4%
- SB204 8% or 12 % (Experimental): SB204 8 or 12 % (supratherapeutic) once
  Interventions: Drug: SB204 8% or 12%
- Moxifloxacillin (No Intervention): Moxifloxacillin 400 mg orally
- Vehicle Gel (Placebo Comparator): Placebo
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SB204 4% — Applied topically once
  Other Names: NVN1000
  Arms: SB204 4%
Drug: SB204 8% or 12% — Applied once topically
  Other Names: NVN1000
  Arms: SB204 8% or 12 %
Drug: Vehicle — Applied topically once
  Other Names: Placebo
  Arms: Vehicle Gel

SUMMARY:
A Double-Blind, Double-Dummy, Randomized, 4-Period Crossover Study to Define the ECG Effects of SB204 Using a Clinical and Supratherapeutic Dose Compared with Placebo and Moxifloxacin (a Positive Control) in Subjects with Acne Vulgaris: A Thorough ECG Study

DETAILED DESCRIPTION:
A Double-Blind, Double-Dummy, Randomized, 4-Period, Crossover Study to Define the ECG Effects of SB204 Using a Clinical and a Supratherapeutic Dose Compared with Placebo and Moxifloxacin (a Positive Control) in Subjects with Acne Vulgaris: A Thorough ECG Study

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe acne
* 20 inflammatory and 25 non-inflammatory acne lesions

Exclusion Criteria:

* Pregnant, trying to become pregnant, or nursing
* Known allergy to any component of the topical SB204 formulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Define ECG effect of SB204 at therapeutic and supratherapeutic dose concentrations as measured by the difference between time-matched baseline adjusted QTcF interval for the groups recieving SB204 and placebo. | 15 days

SECONDARY OUTCOMES:
Categorical analysis of the QTc interval to determine number and percentage of time points and subjects by dose group with absolute QT/QTc > 450, 480, and 500 ms. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, MD, Principal Investigator — Novan, Inc.
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No